CLINICAL TRIAL: NCT06136897
Title: MATCH Treatment Subprotocol J: Trastuzumab and Pertuzumab (HP) in Patients With Non-Breast, Non-Gastric/GEJ, and Non-Colorectal Cancers With HER2 Amplification
Brief Title: Testing Trastuzumab and Pertuzumab in Patients With Higher Than Normal Copies of the HER2 Gene Found in Their Tumors (MATCH - Subprotocol J)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-09506; NCI-2023-09506 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-J (Other: ECOG-ACRIN Cancer Research Group); EAY131-J (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Biopsy; Specimen Handling; pertuzumab; 2C4 antibody; X-Rays; Trastuzumab; CT-P6; PF-05280014; trastuzumab biosimilar HLX02; Ogivri; Ontruzant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pertuzumab, trastuzumab) (Experimental): Patients receive pertuzumab IV over 30-60 minutes and trastuzumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo radiologic evaluation throughout the trial, ECHO at screening and end of treatment, and biopsy and collection of blood samples on trial and at end of treatment.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Biological: Pertuzumab; Procedure: Radiologic Examination; Biological: Trastuzumab

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Biological: Pertuzumab — Given IV
  Other Names: 2C4; 2C4 Antibody; BCD-178; EG1206A; HLX11; HS627; MoAb 2C4; Monoclonal Antibody 2C4; Omnitarg; Perjeta; Pertuzumab Biosimilar BCD-178; Pertuzumab Biosimilar EG1206A; Pertuzumab Biosimilar HLX11; Pertuzumab Biosimilar HS627; Pertuzumab Biosimilar TQB2440; Rhumab 2C4; rhuMAb2C4; RO4368451; TQB 2440; TQB-2440; TQB2440
Procedure: Radiologic Examination — Undergo radiologic evaluation
  Other Names: Radiologic Evaluation; Radiologic Exam
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Biceltis; CANMab; CT-P06; CT-P6; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Hercessi; Herclon; Hertraz; Herwenda; Herzuma; HLX 02; HLX-02; HLX02; Kanjinti; Ogivri; Ontruzant; PF 05280014; PF-05280014; PF05280014; QL 1701; QL-1701; QL1701; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; Trastuzumab Biosimilar CT-P6; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar QL1701; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-herw; Trastuzumab-pkrb; Trastuzumab-qyyp; Trastuzumab-strf; Trastuzumab-zerc; Trazimera; Zercepac

SUMMARY:
This phase II MATCH treatment trial tests how well trastuzumab and pertuzumab work in treating patients with HER2-amplified non-breast, non-gastric/gastroesophageal junction, and non-colorectal cancers. Pertuzumab and trastuzumab are monoclonal antibodies and forms of targeted therapy that attach to a receptor protein called HER2. HER2 is found on some cancer cells. When pertuzumab or trastuzumab attach to HER2, the signals that tell the cells to grow are blocked and the tumor cell may be marked for destruction by the body's immune system. Trastuzumab is approved for the treatment of certain types of HER2-amplified cancers such as breast and gastric cancers. Research has shown that treatment with two anti-HER2 therapies in combination may be more effective at treating HER2-positive patients than giving one anti-HER2 therapy alone. Giving trastuzumab and pertuzumab in combination may be effective at treating patients with HER2-amplified cancers that aren't breast, gastric, or colorectal.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive pertuzumab intravenously (IV) over 30-60 minutes and trastuzumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo radiologic evaluation throughout the trial, echocardiography (ECHO) at screening and end of treatment, and biopsy and collection of blood samples on trial and at end of treatment.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 1 year.

THE MATCH SCREENING TRIAL:

Please see NCT02465060 for information on the MATCH Screening Protocol and applicable documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol
* Patients must fulfill all eligibility criteria outlined the MATCH Master Protocol at the time of registration to treatment step (step 1, 3, 5, 7)
* Patients must have HER2 amplification, or another aberration, as determined via the MATCH Master Protocol
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients must have ECHO or multigated acquisition scan (MUGA) within 4 weeks prior to treatment assignment and must not have a left ventricular ejection fraction (LVEF) < institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be >= 50% for the patient to be eligible
* Patients must not have breast cancer, gastric/gastroesophageal junction (GEJ)/esophageal adenocarcinoma or mixed histology, gastric/GEJ not otherwise specified (NOS) tumors, or colorectal adenocarcinoma
* Patients must not have known hypersensitivity to trastuzumab or pertuzumab or compounds of similar chemical or biologic composition
* Patients must not have received prior anti-HER2 therapies, including trastuzumab, pertuzumab, trastuzumab emtansine (T-DM1), lapatinib, afatinib, neratinib, dacomitinib, canertinib
* Women of childbearing potential (WOCBP) and men who are sexually active with WOCBP must agree to use adequate contraception (hormonal or double barrier method of birth control, abstinence) from one week prior to study treatment starting, during treatment, and for a period of 7 months after the last dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Roisin M Connolly, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Connolly RM, Wang V, Hyman DM, Grivas P, Mitchell EP, Wright JJ, Sharon E, Gray RJ, McShane LM, Rubinstein LV, Patton DR, Williams PM, Hamilton SR, Wang J, Wisinski KB, Tricoli JV, Conley BA, Harris LN, Arteaga CL, O'Dwyer PJ, Chen AP, Flaherty KT. Trastuzumab and Pertuzumab in Patients with Non-Breast/Gastroesophageal HER2-Amplified Tumors: Results from the NCI-MATCH ECOG-ACRIN Trial (EAY131) Subprotocol J. Clin Cancer Res. 2024 Apr 1;30(7):1273-1280. doi: 10.1158/1078-0432.CCR-23-0633. PMID 38433347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol J was activated on March 13, 2017. Thirty-five patients were enrolled between March 2017 and June 2019. Eleven patients were enrolled on the basis of the results from the NCI-MATCH assay and 24 on the basis of the outside assay results.
Pre-assignment Details: Patients with HER2 amplification as established in the analytical assay (CN ≥7) detected by NGS, were considered for the Arm J subprotocol. The mutation status was determined by an NCI-MATCH approved laboratory for 24 patients in this arm, these cases had to be confirmed to be used in primary analysis.
Groups:
- Treatment (Pertuzumab, Trastuzumab): Patients receive pertuzumab IV over 30-60 minutes and trastuzumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Pertuzumab was administered before trastuzumab each cycle; 840 mg loading dose and 420 mg thereafter. Trastuzumab loading dose was 8 mg/kg then 6 mg/kg thereafter. Patients also undergo radiologic evaluation throughout the trial, ECHO at screening and end of treatment, and biopsy and collection of blood samples on trial and at end of treatment.
Period: Overall Study
Arm/Group | Treatment (Pertuzumab, Trastuzumab)
Started | 35
Started Protocol Therapy | 35
Eligible and Treated | 32
Eligible, Treated and Mutation Status Confirmed (Primary efficacy analysis set) | 25
Completed | 0
Not Completed | 35
Not completed — Ineligible | 3
Not completed — Mutation status not confirmed | 7
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Disease progression | 18
Not completed — Other complicating disease | 1
Not completed — Withdrawal by Subject | 1
Not completed — Still on treatment | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Patients who were eligible, started protocol therapy, and had mutation status confirmed at the analysis time were the analyzable patients
Arm/Group | Treatment (Pertuzumab, Trastuzumab)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 66 [31 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Details about how to define complete response and partial response can be found in the master protocol. 90% two-sided binomial exact confidence interval is calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 3 cycles for the first 33 cycles, and every 4 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pertuzumab, Trastuzumab)
Number analyzed (Participants) | 25
percentage of participants | 12 [3.4 to 28.2]

2. Secondary Outcome: 6-month Progression-Free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: as for outcome 1
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pertuzumab, Trastuzumab)
Number analyzed (Participants) | 25
percentage of participants | 25.3 [10.7 to 40]

3. Secondary Outcome: Progression Free Survival
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: as for outcome 1
Population: Eligible, treated and mutation status confirmed
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Pertuzumab, Trastuzumab)
Number analyzed (Participants) | 25
months | 3.3 [2 to 4.1]

ADVERSE EVENTS:
Time Frame: Assessed every 21 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All 35 patients were included in the all-cause mortality and toxicity analysis.
Arm/Group | Treatment (Pertuzumab, Trastuzumab)
All-Cause Mortality (participants affected / at risk) | 27/35
Serious Adverse Events (participants affected / at risk) | 9/35
Other Adverse Events (participants affected / at risk) | 27/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pertuzumab, Trastuzumab) (N=35)
Heart failure (Cardiac disorders) | 2
Fatigue (General disorders) | 1
Infusion related reaction (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Alkaline phosphatase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Stroke (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pertuzumab, Trastuzumab) (N=35)
Anemia (Blood and lymphatic system disorders) | 5
Sinus tachycardia (Cardiac disorders) | 2
Chills (General disorders) | 4
Fatigue (General disorders) | 7
Fever (General disorders) | 2
Infusion related reaction (General disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 3
Weight loss (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT06136897/Prot_001.pdf